CLINICAL TRIAL: NCT02330341
Title: Effect of Artemisia Dracunculus on Glucose Intolerance, Insulin Sensitivity and Insulin Secretion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Manuel González Ortiz, Researcher Professor, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GI-ESTRAGON
Record Dates: First submitted 2014-12-30; First posted 2015-01-01 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Glucose Intolerance
Keywords: Glucose Intolerance; Artemisia dracunculus; Insulin
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: This is a study with two groups of patients with prediabetes. One group received the investigational product (Artemisia Dracunculus) and the other received placebo as control.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artemisia Dracunculus (Experimental): Artemisia Dracunculus extract, 2 capsules of 500 mg, two times per day before breakfast and dinner during 90 days
  Interventions: Dietary Supplement: Artemisia dracunculus
- Placebo (Placebo Comparator): Calcined magnesia, 2 capsules of 500 mg, two times per day before breakfast and dinner during 90 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Artemisia dracunculus
  Other Names: estragon, tarragon
  Arms: Artemisia Dracunculus
Other: Placebo
  Other Names: calcined magnesia
  Arms: Placebo

SUMMARY:
The term prediabetes has been used to encompass the first alterations on glucose metabolism such as impaired fasting glucose and glucose intolerance, and its early detection and treatment could prevent the appearance of diabetes mellitus type 2, a high prevalence disease worldwide.

Artemisia dracunculus, also known as estragon, has been used in Ayurvedic medicine for the treatment of diabetes.

Different in vitro and in vivo studies have shown that Artemisia dracunculus increases insulin signaling and improves insulin sensitivity.

The aim of this study is evaluate the effect of Artemisia dracunculus on glucose intolerance, insulin sensitivity and insulin secretion.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trial will be carried out in 24 patients with diagnosis of glucose intolerance in accordance with the criteria of American Diabetes Association (ADA). Glucose, insulin levels, lipid profile, creatinine, uric acid, and transaminases will be evaluated. An oral glucose tolerance test with 75 g of dextrose will be held.

12 participants will receive Artemisia dracunculus, 1000 mg, twice per day (2000 mg) before breakfast and dinner during 3 months. And other 12 patients will receive placebo with the same prescription.

Area Under de Curve of glucose and insulin will be calculated as well as total insulin secretion (insulinogenic index), first-phase of insulin secretion (Stumvoll index) and insulin sensitivity (Matsuda index).

This protocol is approved by a local ethics committee and written informed consent will be obtained from all volunteers.

Results will be presented as mean and standard deviation. Intra an inter group differences will be tested using the Wilcoxon signed-ran and Mann Whitney U- test respectively; p<0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients both sexes
* Age between 30 and 60 years
* Glucose intolerance according ADA criteria (blood glucose leve ≥140 mg/dl and ≤199 mg/dL after an oral glucose tolerance test with 75 of oral glucose
* Informed consent signed

Exclusion Criteria:

* Women with confirmed or suspected pregnancy
* Women under lactation and/or puerperium
* Hypersensibility to Artemisia dracunculus
* Physical impossibility for taking pills
* Known uncontrolled renal, hepatic, heart or thyroid disease
* Previous treatment for glucose
* Diabetes diagnosis
* BMI ≥39.9 kg/m2

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MANUEL GONZALEZ, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Manuel González Ortiz, Guadalajara, Jalisco, Mexico

RESULTS

PARTICIPANT FLOW:
Groups:
- Artemisia Dracunculus: Artemisia Dracunculus extract, 2 capsules of 500 mg, two times per day before breakfast and dinner during 90 days
  Artemisia dracunculus
- Placebo: Calcined magnesia, 2 capsules of 500 mg, two times per day before breakfast and dinner during 90 days
  Placebo
Period: Overall Study
Arm/Group | Artemisia Dracunculus | Placebo
Started | 12 | 12
Completed | 12 | 11
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Artemisia Dracunculus | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (7) | 48.5 (7.2) | 48.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 24
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 12 | 12 | 24
Postprandial glucose levels [Mean (Standard Deviation); unit: mmol/L] | 10 (1.3) | 9.7 (1.1) | 9.9 (1.2)
Fasting glucose levels [Mean (Standard Deviation); unit: mmol/L] | 5.5 (0.8) | 5.9 (0.9) | 5.7 (0.8)
Glycosylated Hemoglobin [Mean (Standard Deviation); unit: percentage] | 5.8 (0.3) | 5.9 (0.4) | 5.8 (0.4)
First phase of insulin secretion [Mean (Standard Deviation); unit: index] — Human studies support the critical physiologic role of the first-phase of insulin secretion in the maintenance of postmeal glucose homeostasis.
  First phase of insulin secretion was estimated using the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0'), the entered values reflect the first phase of insulin secretion
  index | 1057 (529) | 1395 (1138) | 1226 (885)
Total insulin secretion [Mean (Standard Deviation); unit: index] — The insulinogenic index is a ratio that relates enhancement of circulating insulin to the magnitude of the corresponding glycemic stimulus.
  Total insulin secretion was calculated with the insulinogenic index (ΔABC insulin/ΔABC glucose), the entered values reflect the total insulin secretion
  index | 0.5 (0.2) | 0.7 (0.4) | 0.6 (0.3)
Insulin sensitivity [Mean (Standard Deviation); unit: index] — Matsuda Index value is used to indicate insulin resistance on diabetes. Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]. The entered values reflect the insulin sensitivity
  index | 2.6 (1.3) | 1.9 (1.2) | 2.3 (1.3)
Weight [Mean (Standard Deviation); unit: kilograms] | 85.3 (7.7) | 83 (10.2) | 84.1 (8.9)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 33.1 (2.9) | 34.1 (3.2) | 33.6 (3.0)
Total Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 5.6 (1) | 5 (0.8) | 5.3 (1)
Triglycerides [Mean (Standard Deviation); unit: mmol/L] | 2.5 (1.5) | 1.7 (0.8) | 2.2 (1.3)
High Density Lipoprotein (HDL-c) [Mean (Standard Deviation); unit: mmol/L] | 1.3 (0.3) | 1.4 (0.4) | 1.3 (0.3)
Alanine Aminotransferase (ALT) [Mean (Standard Deviation); unit: U/L] | 43.8 (25.2) | 28.8 (14.1) | 36.3 (21.4)
Aspartate Aminotransferase (AST) [Mean (Standard Deviation); unit: U/L] | 32.2 (17.7) | 26.4 (7.8) | 29.3 (11.3)
Creatinine [Mean (Standard Deviation); unit: umol/L] | 63.7 (8.8) | 65.4 (17.7) | 64.6 (11.5)
Uric Acid [Mean (Standard Deviation); unit: umol/L] | 285.5 (113) | 273.6 (58.9) | 279.6 (132.6)
Systolic blood Pressure [Mean (Standard Deviation); unit: mmHg] | 120 (11) | 123 (10) | 121.6 (10.8)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 78 (7) | 75 (7) | 76.4 (7.5)

OUTCOME MEASURES:

1. Primary Outcome: Postprandial Glucose Levels at Week 12
Description: Postprandial glucose will be evaluated at baseline and week 12 after a oral glucose tolerance test with enzymatic-colorimetric techniques
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Artemisia Dracunculus | Placebo
Number analyzed (Participants) | 12 | 11
mmol/L | 9.5 (1.8) | 9.9 (2.5)
Statistical Analysis 1: Comparison: Artemisia Dracunculus; Results showed in this section are the result of the differences between baseline and final values of postprandial glucose on Artemisia Dracunculus group; Test type: Superiority; p = 0.380, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of postprandial glucose on placebo group; Test type: Superiority; p = 0.695, Wilcoxon (Mann-Whitney); The threshold for statistical significance was p=0.05

2. Primary Outcome: Fasting Glucose Levels at Week 12
Description: Fasting glucose will be evaluated at baseline and week 12 with enzymatic-colorimetric techniques
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Artemisia Dracunculus | Placebo
Number analyzed (Participants) | 12 | 11
mmol/L | 5.9 (0.6) | 5.9 (0.6)
Statistical Analysis 1: Comparison: Artemisia Dracunculus; Results showed in this section are the result of the differences between baseline and final values of fasting glucose on Artemisia Dracunculus group; Test type: Superiority; p = 0.110, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of fasting glucose on placebo group; Test type: Superiority; p = 0.910, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

3. Primary Outcome: Glycosylated Hemoglobin at Week 12
Description: Glycosylated hemoglobin will be evaluated at baseline and week 12 by ELISA
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Artemisia Dracunculus | Placebo
Number analyzed (Participants) | 12 | 11
percentage | 5.6 (0.4) | 5.8 (0.4)
Statistical Analysis 1: Comparison: Artemisia Dracunculus; Results showed in this section are the result of the differences between baseline and final values of glucosylated hemoglobin on Artemisia Dracunculus group; Test type: Superiority; p = 0.010, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of glucosylated hemoglobin on placebo group; Test type: Superiority; p = 0.938, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

4. Primary Outcome: First Phase of Insulin Secretion at Week 12
Description: The first phase of insulin secretion will be calculated at baseline and week 12 with Stumvoll index.
  Human studies support the critical physiologic role of the first-phase of insulin secretion in the maintenance of postmeal glucose homeostasis.
  First phase of insulin secretion was estimated using the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0'), the entered values reflect the first phase of insulin secretion
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Artemisia Dracunculus | Placebo
Number analyzed (Participants) | 12 | 11
index | 1235 (1047) | 1566 (1206)
Statistical Analysis 1: Comparison: Artemisia Dracunculus; Results showed in this section are the result of the differences between baseline and final values of first phase of insulin secretion on Artemisia Dracunculus group; Test type: Superiority; p = 0.733, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of first phase of insulin secretion on placebo group; Test type: Superiority; p = 1.0, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

5. Primary Outcome: Total Insulin Secretion at Week 12
Description: Total insulin secretion will be calculated at baseline and week 12 with insulinogenic index.
  The insulinogenic index is a ratio that relates enhancement of circulating insulin to the magnitude of the corresponding glycemic stimulus.
  Total insulin secretion was calculated with the insulinogenic index (ΔABC insulin/ΔABC glucose), the entered values reflect the total insulin secretion
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Artemisia Dracunculus | Placebo
Number analyzed (Participants) | 12 | 11
index | 0.35 (0.2) | 0.75 (0.4)
Statistical Analysis 1: Comparison: Artemisia Dracunculus; Results showed in this section are the result of the differences between baseline and final values of total insulin secretion on Artemisia Dracunculus group; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of total insulin secretion on placebo group; Test type: Superiority; p = 0.900, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

6. Primary Outcome: Insulin Sensitivity at Week 12
Description: Insulin sensitivity will be calculated at baseline and week 12 with Matsuda index.
  Matsuda Index value is used to indicate insulin resistance on diabetes. Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]. The entered values reflect the insulin sensitivity
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Artemisia Dracunculus | Placebo
Number analyzed (Participants) | 12 | 11
index | 2.4 (1.0) | 1.8 (0.9)
Statistical Analysis 1: Comparison: Artemisia Dracunculus; Results showed in this section are the result of the differences between baseline and final values of insulin sensitivity on Artemisia Dracunculus group; Test type: Superiority; p = 0.519, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of insulin sensitivity on placebo group; Test type: Superiority; p = 0.922, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

7. Secondary Outcome: Weight at Week 12
Description: The weight will be measured at baseline and week 12 with a bioimpedance balance
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Artemisia Dracunculus | Placebo
Number analyzed (Participants) | 12 | 11
kilograms | 85.3 (8.2) | 84.0 (11.0)
Statistical Analysis 1: Comparison: Artemisia Dracunculus; Results showed in this section are the result of the differences between baseline and final values of weight on Artemisia Dracunculus group; Test type: Superiority; p = 0.605, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of weight on placebo group; Test type: Superiority; p = 0.105, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

8. Secondary Outcome: Body Mass Index at Week 12
Description: Body Mass Index will be calculated at baseline and week 12 with the Quetelet index formula
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Artemisia Dracunculus | Placebo
Number analyzed (Participants) | 12 | 11
kg/m^2 | 33.2 (2.9) | 34.4 (3.3)
Statistical Analysis 1: Comparison: Artemisia Dracunculus; Results showed in this section are the result of the differences between baseline and final values of BMI on Artemisia Dracunculus group; Test type: Superiority; p = 0.687, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of BMI on placebo group; Test type: Superiority; p = 0.021, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

9. Secondary Outcome: Total Cholesterol at Week 12
Description: Total cholesterol levels will be evaluated at baseline and week 12 by enzymatic-colorimetric techniques
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Artemisia Dracunculus | Placebo
Number analyzed (Participants) | 12 | 11
mmol/L | 5.4 (1.2) | 5.0 (0.8)
Statistical Analysis 1: Comparison: Artemisia Dracunculus; Results showed in this section are the result of the differences between baseline and final values of total cholesterol on Artemisia Dracunculus group; Test type: Superiority; p = 0.339, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of total cholesterol on placebo group; Test type: Superiority; p = 0.246, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

10. Secondary Outcome: Triglycerides Levels at Week 12
Description: Triglycerides levels will be evaluated at baseline and week 12 with enzymatic-colorimetric techniques
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Artemisia Dracunculus | Placebo
Number analyzed (Participants) | 12 | 11
mmol/L | 2.2 (0.7) | 1.8 (0.9)
Statistical Analysis 1: Comparison: Artemisia Dracunculus; Results showed in this section are the result of the differences between baseline and final values of triglycerides on Artemisia Dracunculus group; Test type: Superiority; p = 0.775, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of triglycerides on placebo group; Test type: Superiority; p = 0.195, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

11. Secondary Outcome: High Density Lipoprotein (c-HDL) Levels at Week 12
Description: c-HDL levels will be evaluated at baseline and week 12 with enzymatic-colorimetric techniques
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Artemisia Dracunculus | Placebo
Number analyzed (Participants) | 12 | 11
mmol/L | 1.4 (0.3) | 1.3 (0.4)
Statistical Analysis 1: Comparison: Artemisia Dracunculus; Results showed in this section are the result of the differences between baseline and final values of HDL-c on Artemisia Dracunculus group; Test type: Superiority; p = 0.040, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of HDL-c on placebo group; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

12. Secondary Outcome: Alanine Aminotransferase (ALT) Levels at Week 12
Description: ALT levels will be evaluated at baseline and week 12 with enzymatic-colorimetric techniques
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Artemisia Dracunculus | Placebo
Number analyzed (Participants) | 12 | 11
U/L | 32.8 (17.7) | 36.7 (18.2)
Statistical Analysis 1: Comparison: Artemisia Dracunculus; Results showed in this section are the result of the differences between baseline and final values of ALT on Artemisia Dracunculus group; Test type: Superiority; p = 0.021, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of ALT on placebo group; Test type: Superiority; p = 0.080, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

13. Secondary Outcome: Aspartate Aminotransferase (AST) Levels at Week 12
Description: AST levels will be evaluated at baseline and week 12 with enzymatic-colorimetric techniques
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Artemisia Dracunculus | Placebo
Number analyzed (Participants) | 12 | 11
U/L | 30.3 (18.1) | 26.7 (9.8)
Statistical Analysis 1: Comparison: Artemisia Dracunculus; Results showed in this section are the result of the differences between baseline and final values of AST on Artemisia Dracunculus group; Test type: Superiority; p = 0.465, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of AST on placebo group; Test type: Superiority; p = 0.574, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

14. Secondary Outcome: Creatinine Levels at Week 12
Description: Creatinine levels will be evaluated at baseline and week 12 with enzymatic-colorimetric techniques
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Artemisia Dracunculus | Placebo
Number analyzed (Participants) | 12 | 11
umol/L | 61.01 (16.8) | 61.01 (13.3)
Statistical Analysis 1: Comparison: Artemisia Dracunculus; Results showed in this section are the result of the differences between baseline and final values of creatinine on Artemisia Dracunculus group; Test type: Superiority; p = 0.480, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of creatinine on placebo group; Test type: Superiority; p = 0.383, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

15. Secondary Outcome: Uric Acid Levels at Week 12
Description: Uric acid levels will be evaluated at baseline and week 12 with enzymatic-colorimetric techniques
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Artemisia Dracunculus | Placebo
Number analyzed (Participants) | 12 | 11
umol/L | 350.9 (71.4) | 309.3 (50.6)
Statistical Analysis 1: Comparison: Artemisia Dracunculus; Results showed in this section are the result of the differences between baseline and final values of uric acid on Artemisia Dracunculus group; Test type: Superiority; p = 0.034, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of uric acid on placebo group; Test type: Superiority; p = 0.080, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

16. Secondary Outcome: Systolic Blood Pressure at Week 12
Description: Systolic blood pressure will be measured at baseline and week 12 with a digital sphygmomanometer
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Artemisia Dracunculus | Placebo
Number analyzed (Participants) | 12 | 11
mmHg | 113 (11) | 125 (8)
Statistical Analysis 1: Comparison: Artemisia Dracunculus; Results showed in this section are the result of the differences between baseline and final values of systolic blood pressure on Artemisia Dracunculus group; Test type: Superiority; p = 0.017, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of systolic blood pressure on placebo group; Test type: Superiority; p = 0.082, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

17. Secondary Outcome: Diastolic Blood Pressure at Week 12.
Description: Diastolic blood pressure will be measured at baseline and week 12 with a digital sphygmomanometer
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Artemisia Dracunculus | Placebo
Number analyzed (Participants) | 12 | 11
mmHg | 75 (8) | 79 (9)
Statistical Analysis 1: Comparison: Artemisia Dracunculus; Results showed in this section are the result of the differences between baseline and final values of diastolic blood pressure on Artemisia Dracunculus group; Test type: Superiority; p = 0.170, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of diastolic blood pressure placebo group; Test type: Superiority; p = 0.199, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 12 weeks of the study.
Arm/Group | Artemisia Dracunculus | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Artemisia Dracunculus (N=12) | Placebo (N=12)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes